CLINICAL TRIAL: NCT01316887
Title: A 52 Week Study to Evaluate the Safety and Tolerability of GSK573719/GW642444 125mcg Once-daily Alone and in Combination With GW642444 25mcg Once-daily Via Novel Dry Powder Inhaler (nDPI) in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A 52-Week, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Safety and Tolerability of GSK573719/GW642444 and GSK573719 in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPD nDPI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 113359
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD; nDPI; long-acting beta agonist; long-acting muscarinic antagonist; tolerability; safety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK573719/GW642444 (Experimental): 125/25 mcg once-daily
  Interventions: Drug: 125/25 mcg once-daily GSK573719/GW642444
- GSK573719 (Experimental): 125 mcg once-daily
  Interventions: Drug: 125mcg once-daily GSK573719
- Placebo (Placebo Comparator): inactive
  Interventions: Drug: Placebo once-daily

INTERVENTIONS:
Drug: 125/25 mcg once-daily GSK573719/GW642444 — GSK573719/GW642444
  Arms: GSK573719/GW642444
Drug: 125mcg once-daily GSK573719 — GSK573719
  Arms: GSK573719
Drug: Placebo once-daily — inactive
  Arms: Placebo

SUMMARY:
The purpose of this 52-week study is to evaluate the long-term safety (in terms of adverse events, COPD exacerbations, laboratory, ECG, and Holter findings, vital signs, use of rescue medication and lung function) of GSK573719/GW642444 Inhalation Powder 125/25mcg in subjects with COPD. The long-term safety of GSK573719 Inhalation Powder 125mcg will also be evaluated. A placebo arm is included to evaluate these products compared to an inactive control.

DETAILED DESCRIPTION:
Several studies have demonstrated the efficacy and safety of combining an individual LABA compound plus an individual LAMA compound in COPD. These studies have shown the combination of these two products to be superior to either agent alone on a variety of outcomes in COPD. The beneficial effects of this combination regimen are likely due to the different mechanisms of action of the two bronchodilators (smooth bronchial muscle relaxation from activation of beta2 receptors from the LABA product and inhibition of acetylcholine-mediated smooth bronchial muscle contraction via blockade of muscarinic receptors from the LAMA product). The availability of a LABA/LAMA combination in one product instead of two individual products is a technical and therapeutic advancement in the pharmacological armamentarium for COPD and may lead to increased patient compliance due to once-daily administration. The purpose of this 52-week study is to evaluate the long-term safety (in terms of adverse events, COPD exacerbations, laboratory, ECG, and Holter findings, vital signs, use of rescue medication, and lung function) of GSK573719/GW642444 Inhalation Powder 125/25mcg in subjects with COPD. The long-term safety of GSK573719 Inhalation Powder 125mcg will also be evaluated. A placebo arm is included to evaluate these products compared to an inactive control. All treatments will be delivered once-daily via the nDPI. This study will establish the long-term safety profile of GSK573719/GW642444 Inhalation Powder 125/25mcg once-daily in subjects with COPD. The safety profile of GSK573719 Inhalation Powder125mcg once-daily will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* outpatient
* signed and dated written informed consent
* 40 years of age or older
* male and female subjects
* COPD diagnosis
* at least 10 pack-year smoking history
* post-albuterol/salbutamol FEV1/FVC ratio of <0.70 and post-albuterol/salbutamol FEV1 greater than or equal to 35% and less than or equal to 80% of predicted normal

Exclusion Criteria:

* Pregant or lactating women or women planning to become pregnant during the study
* current diagnosis of asthma
* other respiratory disorders other than COPD
* other diseases/abnormalities that are uncontrolled including cancer not in remission for at least 5 years
* chest x-ray or CT scan with clinically significant abnormalities not believed to be due to COPD
* hypersensitivity to anticholinergics, beta-agonists, lactose/milk protein or magnesium stearate or medical conditions associated with inhaled anticholinergics
* hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1
* lung volume reduction surgery within 12 months prior to Visit 1
* abnormal and clinically significant ECG at Visit 1
* abnormal and clinically significant Holter monitor finding at Visit 1
* significantly abnormal finding from laboratory tests at Visit 1
* unable to withhold albuterol/salbutamol and/or ipratropium bromide at least 4 hours prior to spirometry at each visit
* use of depot corticosteroids within 12 weeks of Visit 1
* use of oral or parenteral corticosteroids within 6 weeks of Visit 1
* use of anitbiotics for lower respiratory tract infection within 6 weeks of Visit 1
* use of cytochrome P450 3A4 inhibitors within 6 weeks of Visit 1
* us of long-acting beta-agonist (LABA)/inhaled corticosteroid (ICS) products if LABA/ICS therapy is discontinued completely within 30 days of Visit 1
* use of ICS at a dose of >10000mcg/day of fluticasone propionate or equivalent within 30 days of Visit 1
* initiation or discontinuation of ICS within 30 days of Visit 1
* use of tiotropium within 14 days of Visit 1
* use of roflumilast within 14 days of Visit 1
* use of theophyllines within 48 hours of Visit 1
* use of oral leukotriene inhibitors within 48 hours prior to Visit 1
* use of long-acting oral beta-agonists within 48 hours of Visit 1
* use of short-acting oral beta-agonists within 12 hours of Visit 1
* use of inhaled long-acting beta-agonists within 48 hours prior to Visit 1
* use of LABA/ICS combination products only if discontinuing LABA therapy and switching to ICS monotherapy within 48 hours of Visit 1 for the LABA component
* use of sodium cromoglycate or nedocromil sodium within 24 hours of Visit 1
* use of inhaled short acting beta-agonists within 4 hours of Visit 1
* use of inhaled short-acting anticholinergics within 4 hours of Visit 1
* use of inhaled short-acting anticholinergic/short-acting beta2-agonist combination products within 4 hours of Visit 1
* use of any other investigational medication within 30 days or 5 drug half-lives (whichever is longer) of Visit 1
* long-term oxygen therapy prescribed for >12 hours per day
* regular use of short-acting bronchodilators
* use of CPAP or NIPPV
* participation in the maintenance phase of a pulmonary rehabilitation program
* known or suspected history of alcohol or drug abluse with 2 years prior to Visit 1
* anyone affiliated with the investigator site (e.g., investigator, study coordinator, etc.)
* previous use of GSK573719, GW642444 , GSK573719/GW642444 combination, GSK233705/GW642444 combination, or Fluticasone Furoate/GW642444 combination

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2011-01-01; Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (15):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Morgantown, West Virginia
- Chile (3):
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Talca, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Romania (6):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Timișoara
- Russia (12):
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Penza
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Shakhty, Rostov Region
  - GSK Investigational Site, Sochi
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Tyumen
  - GSK Investigational Site, Veliky Novgorod
  - GSK Investigational Site, Vladivostok
  - GSK Investigational Site, Yekaterinburg
- Slovakia (5):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Poprad
  - GSK Investigational Site, Považská Bystrica
  - GSK Investigational Site, Šaľa
  - GSK Investigational Site, Žilina
- South Africa (8):
  - GSK Investigational Site, Benoni, Gauteng
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Gatesville
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Tygerberg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 113359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a Run-in Period of 7 to10 days, followed by a 52-week Treatment Period. A total of 893 participants were screened; of these, 312 were screen failures, 19 were Run-in failures, 563 were randomized, and 562 received at least one dose of study drug (one participant was randomized in error but did not receive study drug).
Groups:
- Placebo: Participants received matching placebo once daily (QD) in the morning via a dry powder inhaler (DPI) for 52 weeks.
- UMEC 125 µg: Participants received umeclidinium bromide (UMEC) 125 micrograms (µg) QD in the morning via a DPI for 52 weeks.
- UMEC/VI 125/25 µg: Participants received umeclidinium bromide/vilanterol (UMEC/VI) 125/25 µg QD in the morning via a DPI for 52 weeks.
Period: Overall Study
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Started | 109 | 227 | 226
Completed | 66 | 133 | 143
Not Completed | 43 | 94 | 83
Not completed — Adverse Event | 13 | 21 | 17
Not completed — Lack of Efficacy | 9 | 3 | 1
Not completed — Protocol Violation | 2 | 6 | 6
Not completed — Protocol-defined Stopping Criteria | 8 | 37 | 36
Not completed — Study Closed/Terminated | 2 | 4 | 3
Not completed — Lost to Follow-up | 1 | 7 | 5
Not completed — Withdrawal by Subject | 8 | 16 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg | Total
Number analyzed (Participants) | 109 | 227 | 226 | 562
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (8.28) | 61.7 (9.10) | 61.4 (9.01) | 61.3 (8.92)
Sex/Gender, Customized [Number; unit: Participants]
  African American/African Heritage (HER) | 3 | 13 | 14 | 30
  Japanese/East Asian HER/South East Asian HER | 2 | 0 | 1 | 3
  White | 104 | 214 | 211 | 529
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 82 | 70 | 188
  Male | 73 | 145 | 156 | 374

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any On-treatment Adverse Event (AE) or Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury with hyperbilirubinaemia. Medical or scientific judgment was to have been exercised in other important medical events. AEs with an onset on or after the date of the first dose of study drug and up to 1 day after the date of the last recorded dose of study drug were considered to be on-treatment AEs, Refer to the general AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the start of study drug up to 52 weeks
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of randomized study drug
Measure: Number; unit: Participants
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
Participants
  Any on-treatment AE | 57 | 132 | 120
  Any on-treatment SAE | 7 | 17 | 14

2. Secondary Outcome: Number of Participants With at Least One Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Over the Course of the 52-week Treatment Period
Description: A COPD exacerbation is defined as worsening symptoms of COPD requiring a systemic corticosteroid, an antibiotic, and/or hospitalization.
Time Frame: From the start of study drug up to 52 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
Participants | 26 | 33 | 29

3. Secondary Outcome: Time to the First On-treatment COPD Exacerbation
Description: An on-treatment COPD exacerbation is defined as worsening symptoms of COPD requiring a systemic corticosteroid, an antibiotic, and/or hospitalization at any time during the 52-week Treatment Period. The time to the first on-treatment exacerbation was calculated as the exacerbation onset date of the first on-treatment exacerbation minus the date of the start of treatment + 1. The median time to the first on-treatment exacerbation was derived from the Kaplan-Meier analysis. A participant who did not experience an exacerbation prior to completing the study or withdrawal is considered censored; a time to first COPD exacerbation cannot be calculated for these participants.
Time Frame: From the start of study drug up to 52 weeks
Population: ITT Population
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
Days | NA [1 to 372] — Per Kaplan-Meier analysis, because 50% of the data were censored, the median could not be calculated. | NA [1 to 372] — Per Kaplan-Meier analysis, because 50% of the data were censored, the median could not be calculated. | NA [1 to 372] — Per Kaplan-Meier analysis, because 50% of the data were censored, the median could not be calculated.

4. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Creatine Kinase (CK), and Gamma Glutamyl Transferase (GGT) at Months 3, 6, 9, and 12
Description: Blood samples were collected for the measurement of ALT, ALP, AST, CK, and GGT at Baseline and Months 3, 6, 9, and 12. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The value defined as the "Baseline" value is the most recent value collected prior to the start of treatment. For most participants, the Baseline value is the value collected at the Screening visit; however, for some participants, the Baseline value may have been collected at an unscheduled visit.
Time Frame: Baseline; Months 3, 6, 9, and 12
Population: ITT Population. Only those participants available at the specified time points were summarized (represented by n=X, X, X in the category titles). Different participants may have been summarized for different parameters/at different time points, so the overall number of participants summarized reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
International units per liter (IU/L)
  ALT, Month 3, n=88, 190, 193 | 0.3 (12.53) | 0.8 (9.40) | 0.6 (15.27)
  ALT, Month 6, n=73, 158, 172 | -1.3 (14.03) | 3.2 (22.35) | 1.0 (16.83)
  ALT, Month 9, n=69, 148, 149 | -0.6 (12.81) | -0.2 (7.64) | -0.5 (14.68)
  ALT, Month 12, n=65, 129, 140 | -1.7 (14.92) | 1.3 (15.63) | -1.7 (17.53)
  ALP, Month 3, n=88, 190, 193 | 1.1 (21.90) | -1.6 (12.13) | 0.3 (12.91)
  ALP, Month 6, n=73, 158, 172 | -0.4 (23.35) | -1.6 (17.15) | -0.9 (14.44)
  ALP, Month 9, n=69, 148, 149 | -1.5 (18.53) | -2.2 (12.68) | 0.0 (16.51)
  ALP, Month 12, n=65, 129, 140 | -1.9 (18.09) | 4.3 (61.45) | 0.2 (15.93)
  AST, Month 3, n=88, 190, 192 | 0.1 (19.27) | 1.3 (10.87) | 1.0 (14.75)
  AST, Month 6, n=73, 158, 172 | -2.8 (18.52) | 3.8 (23.71) | 1.3 (16.50)
  AST, Month 9, n=69, 148, 148 | -1.1 (10.79) | 0.1 (6.53) | -1.1 (12.95)
  AST, Month 12, n=65, 129, 140 | -0.6 (12.06) | 2.6 (15.71) | -0.8 (12.01)
  CK, Month 3, n=88, 190, 193 | 2.4 (84.76) | -1.8 (97.44) | 7.0 (63.51)
  CK, Month 6, n=73, 158, 172 | -8.3 (41.87) | 3.6 (114.53) | 10.8 (94.52)
  CK, Month 9, n=69, 148, 149 | 3.8 (55.89) | -2.3 (113.58) | 3.5 (58.82)
  CK, Month 12, n=64, 129, 140 | -1.8 (46.31) | 0.9 (118.66) | 16.7 (68.75)
  GGT, Month 3, n=88, 190, 193 | 11.5 (95.98) | 1.0 (24.07) | -2.1 (53.42)
  GGT, Month 6, n=73, 158, 172 | -5.6 (48.15) | 9.8 (73.28) | 1.5 (27.49)
  GGT, Month 9, n=69, 148, 149 | -1.3 (25.59) | -0.5 (22.45) | -2.5 (39.81)
  GGT, Month 12, n=65, 129, 140 | -6.9 (44.77) | 7.8 (72.04) | -2.0 (30.93)

5. Secondary Outcome: Change From Baseline in Albumin, Total Protein, and Hemoglobin at Months 3, 6, 9, and 12
Description: Blood samples were collected for the measurement of albumin, total protein, and hemoglobin at Baseline and Months 3, 6, 9, and 12. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The value defined as the "Baseline" value is the most recent value collected prior to the start of treatment. For most participants, the Baseline value is the value collected at the Screening visit; however, for some participants, the Baseline value may have been collected at an unscheduled visit.
Time Frame: Baseline; Months 3, 6, 9, and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Groups:
- UMEC/VI 125/25µg: Participants received umeclidinium bromide/vilanterol (UMEC/VI) 125/25 µg QD in the morning via a DPI for 52 weeks.
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25µg
Number analyzed (Participants) | 109 | 227 | 226
Grams per liter (G/L)
  Albumin, Month 3, n=88, 190, 193 | -0.5 (2.44) | -0.8 (2.48) | -0.8 (2.67)
  Albumin, Month 6, n=73, 158, 172 | -0.6 (2.89) | -0.9 (2.59) | -0.4 (2.85)
  Albumin, Month 9, n=69, 149, 149 | -0.1 (3.19) | -0.8 (2.55) | -0.5 (3.31)
  Albumin, Month 12, n=65, 129, 140 | -1.2 (3.27) | -1.4 (2.35) | -0.9 (3.00)
  Total protein, Month 3, n=88, 190, 193 | -1.2 (3.99) | -1.3 (3.52) | -1.1 (3.91)
  Total protein, Month 6, n=73, 158, 172 | -1.1 (4.01) | -1.8 (3.57) | -0.7 (4.10)
  Total protein, Month 9, n=69, 148, 149 | -0.7 (4.50) | -1.8 (3.52) | -1.4 (4.56)
  Total protein, Month 12, n=65, 129, 140 | -2.1 (4.48) | -2.6 (3.48) | -1.9 (3.82)
  Hemoglobin, Month 3, n=94, 198, 206 | -1.2 (8.51) | -1.5 (8.05) | -2.0 (8.34)
  Hemoglobin, Month 6, n=75, 159, 171 | -1.6 (9.85) | -1.2 (7.31) | -1.4 (9.31)
  Hemoglobin, Month 9, n=70, 152, 155 | -1.4 (11.95) | -2.5 (10.35) | -2.2 (8.78)
  Hemoglobin, Month 12, n=63, 130, 143 | -2.7 (11.36) | -2.5 (7.04) | -2.1 (9.19)

6. Secondary Outcome: Change From Baseline in Calcium, Carbon Dioxide (CO2) Content/Bicarbonate, Chloride, Glucose, Inorganic Phosphorus (IP), Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) at Months 3, 6, 9, and 12
Description: Blood samples were collected for the measurement of calcium, CO2 content/bicarbonate, chloride, glucose, IP, potassium, sodium, and urea/BUN at Baseline and Months 3, 6, 9, and 12. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The value defined as the "Baseline" value is the most recent value collected prior to the start of treatment. For most participants, the Baseline value is the value collected at the Screening visit; however, for some participants, the Baseline value may have been collected at an unscheduled visit.
Time Frame: Baseline; Months 3, 6, 9, and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
Millimoles per liter (mmol/L)
  Calcium, Month 3, n=88, 189, 192 | -0.004 (0.0957) | -0.006 (0.1178) | -0.016 (0.0990)
  Calcium, Month 6, n=73, 157, 172 | -0.027 (0.0893) | -0.011 (0.1058) | 0.000 (0.1104)
  Calcium, Month 9, n=69, 147, 148 | -0.027 (0.1009) | -0.019 (0.1036) | -0.014 (0.1023)
  Calcium, Month 12, n=65, 129, 140 | -0.023 (0.1070) | -0.007 (0.0959) | -0.009 (0.1059)
  CO2 content/bicarbonate, Month 3, n=88, 190, 192 | 0.8 (2.99) | 0.8 (2.70) | 0.6 (2.87)
  CO2 content/bicarbonate, Month 6, n=73, 158, 172 | 0.3 (3.03) | 0.2 (2.84) | 0.7 (3.14)
  CO2 content/bicarbonate, Month 9, n=69, 149, 148 | 0.3 (3.21) | 0.2 (2.78) | 0.3 (2.87)
  CO2 content/bicarbonate, Month 12, n=65, 129, 140 | -0.6 (3.06) | -0.3 (2.70) | -0.4 (2.49)
  Chloride, Month 3, n=88, 190, 193 | 0.0 (3.03) | -0.2 (3.33) | -0.1 (2.60)
  Chloride, Month 6, n=73, 158, 172 | -0.2 (2.84) | -0.2 (2.90) | -0.1 (3.23)
  Chloride, Month 9, n=69, 149, 149 | -0.7 (3.27) | -0.3 (2.93) | -0.5 (2.94)
  Chloride, Month 12, n=64, 129, 140 | -0.2 (3.08) | 0.0 (2.56) | 0.3 (2.86)
  Glucose, Month 3, n=88, 190, 193 | 0.08 (1.269) | 0.08 (1.315) | 0.03 (1.419)
  Glucose, Month 6, n=73, 158, 172 | 0.22 (1.412) | 0.18 (1.645) | -0.01 (2.507)
  Glucose, Month 9, n=69, 149, 149 | 0.18 (1.333) | 0.16 (1.959) | 0.05 (2.309)
  Glucose, Month 12, n=65, 129, 140 | 0.19 (1.080) | 0.00 (1.741) | 0.01 (2.453)
  IP, Month 3, n=87, 189, 193 | 0.022 (0.1844) | 0.003 (0.1663) | -0.018 (0.1886)
  IP, Month 6, n=72, 157, 171 | 0.016 (0.1880) | 0.015 (0.1686) | 0.027 (0.2125)
  IP, Month 9, n=68, 147, 149 | -0.026 (0.1773) | -0.002 (0.1850) | 0.005 (0.1962)
  IP, Month 12, n=64, 129, 140 | -0.007 (0.1838) | 0.022 (0.1821) | 0.011 (0.1793)
  Potassium, Month 3, n=88, 190, 192 | 0.04 (0.464) | 0.05 (0.490) | 0.08 (0.474)
  Potassium, Month 6, n=73, 158, 171 | -0.05 (0.462) | 0.02 (0.468) | 0.00 (0.428)
  Potassium, Month 9, n=69, 149, 148 | -0.14 (0.461) | -0.01 (0.494) | -0.05 (0.498)
  Potassium, Month 12, n=65, 129, 140 | -0.06 (0.489) | -0.01 (0.473) | -0.04 (0.510)
  Sodium, Month 3, n=88, 190, 193 | -0.1 (2.84) | -0.5 (2.50) | -0.8 (2.36)
  Sodium, Month 6, n=73, 158, 172 | -0.7 (2.31) | -0.8 (2.63) | -0.7 (2.48)
  Sodium, Month 9, n=69, 149, 149 | -0.7 (2.54) | -0.8 (2.72) | -1.0 (2.59)
  Sodium, Month 12, n=64, 129, 140 | -1.0 (2.11) | -0.7 (2.40) | -0.5 (2.75)
  Urea/BUN, Month 3, n=88, 190, 193 | -0.03 (1.961) | -0.18 (1.574) | -0.01 (1.814)
  Urea/BUN, Month 6, n=73, 158, 172 | -0.06 (2.734) | -0.12 (1.698) | 0.00 (1.875)
  Urea/BUN, Month 9, n=69, 149, 149 | -0.12 (1.981) | -0.21 (1.692) | -0.11 (1.696)
  Urea/BUN, Month 12, n=65, 129, 140 | 0.13 (2.591) | -0.29 (1.631) | 0.16 (1.613)

7. Secondary Outcome: Change From Baseline in Creatinine, Direct Bilirubin, Indirect Bilirubin, Total Bilirubin, and Uric Acid at Months 3, 6, 9, and 12
Description: Blood samples were collected for the measurement of creatinine, direct bilirubin, indirect bilirubin, total bilirubin, and uric acid at Baseline and Months 3, 6, 9, and 12. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The value defined as the "Baseline" value is the most recent value collected prior to the start of treatment. For most participants, the Baseline value is the value collected at the Screening visit; however, for some participants, the Baseline value may have been collected at an unscheduled visit.
Time Frame: Baseline; Months 3, 6, 9, and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
Micromoles per liter (µmol/L)
  Creatinine, Month 3, n=88, 190, 193 | -3.20 (16.221) | -1.63 (9.119) | -0.51 (10.034)
  Creatinine, Month 6, n=73, 158, 171 | -0.52 (19.828) | -1.14 (9.047) | 0.13 (11.418)
  Creatinine, Month 9, n=69, 148, 149 | -1.17 (20.543) | -0.71 (9.780) | 0.26 (11.057)
  Creatinine, Month 12, n=65, 129, 140 | -0.06 (20.259) | 1.11 (12.375) | 1.79 (11.571)
  Direct bilirubin, Month 3, n=88, 190, 192 | 0.0 (1.08) | 0.1 (1.13) | 0.0 (1.05)
  Direct Bilirubin, Month 6, n=73, 158, 172 | -0.1 (1.02) | 0.0 (1.20) | 0.0 (0.91)
  Direct bilirubin, Month 9, n=69, 149, 149 | 0.0 (1.06) | -0.2 (0.98) | -0.1 (0.93)
  Direct bilirubin, Month 12, n=65, 129, 139 | 0.1 (0.88) | 0.8 (8.77) | -0.2 (1.12)
  Indirect bilirubin, Month 3, n=88, 190, 192 | 0.1 (3.30) | -0.2 (3.64) | -0.2 (3.03)
  Indirect bilirubin, Month 6, n=73, 158, 172 | -0.1 (3.21) | -0.3 (3.69) | -0.2 (2.94)
  Indirect bilirubin, Month 9, n=69, 148, 149 | 0.2 (3.68) | -0.6 (3.28) | -0.3 (2.93)
  Indirect bilirubin, Month 12, n=65, 129, 139 | -0.2 (2.74) | 0.4 (8.60) | -0.5 (3.51)
  Total bilirubin, Month 3, n=88, 190, 193 | 0.1 (3.76) | 0.0 (4.29) | -0.2 (3.52)
  Total bilirubin, Month 6, n=73, 158, 172 | -0.2 (3.61) | -0.3 (4.37) | -0.2 (3.51)
  Total bilirubin, Month 9, n=69, 148, 149 | 0.2 (4.13) | -0.8 (3.82) | -0.4 (3.41)
  Total bilirubin, Month 12, n=65, 129, 140 | -0.1 (3.06) | 1.2 (17.09) | -0.7 (4.25)
  Uric acid, Month 3, n=88, 189, 193 | -3.4 (68.15) | -0.1 (53.93) | 16.2 (72.11)
  Uric acid, Month 6, n=73, 157, 172 | 2.5 (85.86) | 0.3 (57.74) | 1.9 (63.17)
  Uric acid, Month 9, n=69, 147, 149 | -2.9 (72.40) | -8.3 (61.57) | -1.9 (66.69)
  Uric acid, Month 12, n=65, 129, 140 | 11.4 (80.09) | -2.8 (65.58) | 0.9 (69.74)

8. Secondary Outcome: Change From Baseline in the Percentage of Basophils, Eosinophils, Lymphocytes, Monocytes, and Segmented Neutrophils in Blood at Months 3, 6, 9, and 12
Description: Blood samples were collected for the measurement of the percentage of basophils, eosinophils, lymphocytes, monocytes, and segmented neutrophils at Baseline and Months 3, 6, 9, and 12. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The value defined as the "Baseline" value is the most recent value collected prior to the start of treatment. For most participants, the Baseline value is the value collected at the Screening visit; however, for some participants, the Baseline value may have been collected at an unscheduled visit.
Time Frame: Baseline; Months 3, 6, 9, and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage in blood
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
Percentage in blood
  Basophils, Month 3, n=93, 198, 206 | -0.02 (0.244) | 0.01 (0.290) | 0.02 (0.302)
  Basophils, Month 6, n=73, 156, 167 | -0.03 (0.270) | 0.03 (0.312) | 0.01 (0.314)
  Basophils, Month 9, n=70, 152, 154 | -0.01 (0.265) | 0.02 (0.276) | 0.02 (0.300)
  Basophils, Month 12, n=62, 130, 141 | -0.05 (0.235) | 0.00 (0.240) | 0.02 (0.266)
  Eosinophils, Month 3, n=93, 198, 206 | 0.17 (1.569) | -0.01 (2.243) | -0.05 (1.791)
  Eosinophils, Month 6, n=73, 156, 167 | 0.04 (1.720) | -0.08 (2.101) | 0.27 (1.962)
  Eosinophils, Month 9, n=70, 152, 154 | 0.18 (2.271) | -0.33 (2.232) | 0.02 (1.678)
  Eosinophils, Month 12, n=62, 130, 141 | 0.10 (1.698) | -0.19 (2.557) | 0.09 (2.021)
  Lymphocytes, Month 3, n=93, 198, 206 | -1.02 (8.031) | -1.86 (7.912) | -0.92 (7.474)
  Lymphocytes, Month 6, n=73, 156, 167 | -1.14 (7.178) | -0.33 (10.319) | 0.81 (9.211)
  Lymphocytes, Month 9, n=70, 152, 154 | -2.63 (6.977) | -1.32 (8.439) | -1.35 (8.265)
  Lymphocytes, Month 12, n=62, 130, 141 | -0.93 (6.654) | -0.55 (7.459) | -0.25 (7.138)
  Monocytes, Month 3, n=93, 198, 206 | -0.02 (2.544) | -0.06 (2.303) | 0.13 (2.296)
  Monocytes, Month 6, n=73, 156, 167 | 0.60 (2.929) | 1.09 (3.170) | 0.56 (2.935)
  Monocytes, Month 9, n=70, 152, 154 | 0.14 (2.959) | 0.62 (2.453) | 0.24 (2.466)
  Monocytes, Month 12, n=62, 130, 141 | 0.26 (2.563) | 0.47 (2.632) | -0.16 (2.198)
  Segmented neutrophils, Month 3, n=93, 198, 206 | 0.88 (9.494) | 1.92 (9.714) | 0.81 (9.002)
  Segmented neutrophils, Month 6, n=73, 156, 167 | 0.53 (9.264) | -0.72 (12.744) | -1.65 (11.543)
  Segmented neutrophils, Month 9, n=70, 152, 154 | 2.02 (8.225) | 1.00 (10.311) | 1.07 (9.472)
  Segmented neutrophils, Month 12, n=62, 130, 141 | 0.63 (7.903) | 0.27 (10.026) | 0.29 (8.456)

9. Secondary Outcome: Change From Baseline in Eosinophil Count, Platelet Count, and White Blood Cell (WBC) Count at Months 3, 6, 9, and 12
Description: Blood samples were collected for the measurement of eosinophils, platelets, and WBC count at Baseline and Months 3, 6, 9, and 12. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The value defined as the "Baseline" value is the most recent value collected prior to the start of treatment. For most participants, the Baseline value is the value collected at the Screening visit; however, for some participants, the Baseline value may have been collected at an unscheduled visit.
Time Frame: Baseline; Months 3, 6, 9, and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
10^9 cells per liter (GI/L)
  Eosinophil count, Month 3, n=93, 198, 206 | 0.001 (0.1134) | -0.002 (0.1497) | -0.007 (0.1292)
  Eosinophil count, Month 6, n=73, 156, 167 | -0.005 (0.1246) | -0.007 (0.1277) | 0.015 (0.1324)
  Eosinophil count, Month 9, n=70, 152, 154 | 0.003 (0.1613) | -0.023 (0.1445) | 0.001 (0.1227)
  Eosinophil count, Month 12, n=62, 130, 141 | -0.003 (0.1297) | -0.013 (0.1678) | 0.010 (0.1496)
  Platelet count, Month 3, n=93, 197, 204 | 2.2 (40.22) | -4.4 (38.28) | 4.4 (34.39)
  Platelet count, Month 6, n=73, 155, 169 | -11.6 (39.11) | -5.4 (39.61) | -0.6 (33.65)
  Platelet count, Month 9, n=68, 151, 154 | -9.5 (39.36) | -3.0 (39.85) | 0.7 (37.24)
  Platelet count, Month 12, n=61, 128, 140 | -11.8 (34.45) | -4.4 (33.09) | 4.4 (37.68)
  WBC count, Month 3, n=93, 198, 206 | -0.20 (1.575) | -0.27 (1.781) | -0.21 (1.797)
  WBC count, Month 6, n=73, 156, 167 | -0.06 (1.666) | -0.13 (1.663) | -0.23 (2.065)
  WBC count, Month 9, n=70, 152, 154 | 0.29 (2.820) | -0.09 (1.919) | -0.19 (1.850)
  WBC count, Month 12, n=62, 130, 141 | -0.19 (1.600) | -0.21 (2.114) | -0.09 (1.871)

10. Secondary Outcome: Change From Baseline in Hematocrit at Months 3, 6, 9, and 12
Description: Blood samples were collected for the measurement of hematocrit at Baseline and Months 3, 6, 9, and 12. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The value defined as the "Baseline" value is the most recent value collected prior to the start of treatment. For most participants, the Baseline value is the value collected at the Screening visit; however, for some participants, the Baseline value may have been collected at an unscheduled visit.
Time Frame: Baseline; Months 3, 6, 9, and 12
Population: ITT Population. Only those participants available at the specified time points were summarized (represented by n=X, X, X in the category titles). Different participants may have been summarized at different time points, so the overall number of participants summarized reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
Proportion of red blood cells in blood
  Month 3, n=94, 198, 206 | -0.0140 (0.02757) | -0.0134 (0.02656) | -0.0131 (0.02699)
  Month 6, n=75, 159, 171 | -0.0195 (0.03320) | -0.0177 (0.02446) | -0.0170 (0.02871)
  Month 9, n=70, 152, 155 | -0.0133 (0.03785) | -0.0139 (0.03158) | -0.0146 (0.02829)
  Month 12, n=63, 130, 143 | -0.0072 (0.03336) | -0.0045 (0.02356) | -0.0040 (0.2959)

11. Secondary Outcome: Change From Baseline to Maximum Systolic Blood Pressure (SBP) and Change From Baseline to Minimum Diastolic Blood Pressure (DBP) Over the Course of the 52-week Treatment Period
Description: Baseline is defined as the most recent recorded value before dosing on Day 1. The maximum post-Baseline value for SBP and the minimum post-Basline value for DBP were derived using any scheduled, unscheduled, or early withdrawal visit made after the start of study treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; from the start of study drug up to 52 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
Millimeters of mercury (mmHg)
  Change from Baseline to maximum SBP | 14.5 (15.28) | 14.0 (14.05) | 13.5 (13.02)
  Change from Baseline to minimum DBP | -11.0 (8.87) | -9.5 (7.86) | -10.8 (8.89)

12. Secondary Outcome: Maximum Change From Baseline in Pulse Rate Over the Course of the 52-week Treatment Period
Description: Baseline is defined as the most recent recorded value before dosing on Day 1. The maximum post-Baseline value for pulse rate was derived using any scheduled, unscheduled, or early withdrawal visit made after the start of study treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; from the start of study drug up to 52 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
Beats per minute | 9.1 (9.30) | 9.8 (10.16) | 9.0 (9.04)

13. Secondary Outcome: Maximum Change From Baseline in the Electrocardiogram (ECG) Parameters of QT Interval Corrected for Heart Rate by Bazett's Formula (QTcB), QT Interval Corrected for Heart Rate by Fridericia's Formula (QTcF), and PR Interval Over the Course of the 52-week
Description: 12-lead ECG measurements were obtained. Baseline is defined as the most recent recorded value before dosing on Day 1. The maximum post-Baseline values for QTcF, QTcB, and PR interval were derived using any scheduled, unscheduled, or early withdrawal visit made after the start of study treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; from the start of study drug up to 52 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
Milliseconds
  Maximum change from Baseline in QTcF | 15.6 (13.67) | 16.9 (14.20) | 18.4 (14.42)
  Maximum change from Baseline in QTcB | 17.1 (16.90) | 19.0 (17.62) | 20.7 (17.14)
  Maximum change from Baseline in PR interval | 12.4 (11.03) | 13.5 (10.26) | 12.0 (9.79)

14. Secondary Outcome: Maximum Change From Baseline in the ECG Parameter of Heart Rate Over the Course of the 52-week Treatment Period
Description: 12-lead ECG measurements were obtained. Baseline is defined as the most recent recorded value before dosing on Day 1. The maximum post-Baseline value for heart rate was derived using any scheduled, unscheduled, or early withdrawal visit made after the start of study treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; from the start of study drug up to 52 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
Beats per minute | 7.8 (8.67) | 9.9 (13.66) | 9.3 (9.43)

15. Secondary Outcome: Number of Participants With the Indicated ECG Result Interpretations at Any Time Post-Baseline
Description: Post-Baseline visits include scheduled, unscheduled, and Early Withdrawal visits. Only the worst-case interpretation was counted for each participant. Clinical significance and abnormal/normal findings are based on the assessment of the independent cardiologists.
Time Frame: From the start of study drug up to 52 weeks
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 109 | 227 | 226
participants
  Normal | 32 | 64 | 71
  Abnormal - Not Clinically Significant | 52 | 105 | 101
  Abnormal - Clinically Significant | 25 | 58 | 54
  Unable to Evaluate | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With the Indicated Change From Screening to Any Time Post-Baseline in Holter ECG Interpretation
Description: Twenty-four hour Holter monitor (12-lead) evaluations were obtained. Holter Baseline values were those recorded at Screening. An "any time post-Baseline" Holter evaluation was derived as the worst evaluation recorded at any scheduled, unscheduled, or early withdrawal visit made after the start of study treatment. Change from Screening was calculated as the post-Screening value minus the Screening value. The order of severity for change from Screening Holter evaluation from worst to best is: clinically significant change: unfavorable; no change or insignificant change; clinically significant change: favorable, unable to compare, based on the assessment of the independent cardiologists.
Time Frame: Screening; from the start of study drug up to 52 weeks
Population: ITT Population. Only those participants providing at least one post-Baseline interpretation were summarized.
Measure: Number; unit: Participants
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 90 | 198 | 207
Participants
  Clinically significant change: unfavorable | 39 | 86 | 87
  No change or insignificant change | 46 | 98 | 110
  Clinically significant change: favorable | 3 | 6 | 4
  Unable to compare | 2 | 8 | 6

17. Secondary Outcome: Change From Baseline in the Mean Number of Puffs of Rescue Medication (Salbutamol and/or Ipratropium Bromide) Per Day Over the Course of the 52-week Treatment Period
Description: Participants recorded the number of puffs and/or the number of nebules of rescue albuterol/salbutamol and/or ipratropium bromide used in the past 24 hours for the relief of COPD symptoms in the daily diary. The total puffs of rescue medication for each day was calculated as follows: (number of salbutamol puffs + number of ipratropium puffs + [2 * number of salbutamol nebules] + [2 * number of ipratropium nebules]). Baseline is the mean during the week prior to Day 1. Change from Baseline was calculated as the mean number of puffs/day over Weeks 1-52 minus the mean number of puffs/day at Baseline. Analysis was performed using an Analysis of Covariance (ANCOVA) model with covariates of treatment, Baseline (mean during the week prior to Day 1), smoking status, and center group.
Time Frame: Baseline; from the start of study drug up to 52 weeks
Population: ITT Population. Only those participants who had rescue data available on at least 50% of the days in the 52-week treatment period were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Number of puffs per day
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 75 | 158 | 168
Number of puffs per day | -0.4 (0.20) | -0.8 (0.14) | -1.4 (0.13)

18. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free Days Over the Course of the 52-week Treatment Period
Description: Rescue-free days are defined as days on which albuterol/salbutamol and/or ipratropium bromide was not used. Baseline is the percentage during the week prior to Day 1. Change from Baseline was calculated as the mean percentage of rescue-free days over Weeks 1-52 minus the mean percentage of rescue-free days at Baseline.
Time Frame: From the start of study drug up to 52 weeks
Population: ITT Population. Only those participants who had rescue data available on at least 50% of the days in the 52-week treatment period were included in the summary.
Measure: Mean (Standard Deviation); unit: Percentage of rescue-free days
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 75 | 158 | 168
Percentage of rescue-free days | 11.1 (30.06) | 13.1 (37.35) | 23.2 (39.27)

19. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) and Forced Vital Capacity (FVC) at Months 1, 3, 6, 9, and 12
Description: FEV1 and FVC are measures of lung function. FEV1 is defined as the maximal amount of air that can be forcefully exhaled in one second. FVC is defined as the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. Trough FEV1 and FVC were the values obtained approximately 24 hours after the previous morning's dose of study medication. Baseline is the value recorded pre-dose on Day 1. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Analysis was performed using a repeated measures model with covariates of treatment, Baseline (assessment made immediately pre-dose on Day 1), smoking status, center group, month, and month by Baseline and month by treatment interactions.
Time Frame: Baseline; Months 1, 3, 6, 9, and 12
Population: ITT Population. The overall number of participants reflects all participants who provided at least one post-treatment assessment. Participants who provided data the specified time points are represented by n=X, X, X in the category titles.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Number analyzed (Participants) | 103 | 215 | 216
Liters
  FEV1: Month 1, n=103, 215, 215 | -0.030 (0.0253) | 0.138 (0.0175) | 0.161 (0.0174)
  FEV1: Month 3, n=90, 197, 208 | -0.036 (0.0289) | 0.140 (0.0197) | 0.189 (0.0192)
  FEV1: Month 6, n=79, 163, 178 | -0.015 (0.0320) | 0.144 (0.0221) | 0.181 (0.0214)
  FEV1: Month 9, n=71, 142, 153 | -0.050 (0.0314) | 0.104 (0.0219) | 0.180 (0.0213)
  FEV1: Month 12, n=66, 132, 143 | -0.045 (0.0332) | 0.133 (0.0232) | 0.186 (0.0224)
  FVC: Month 1, n=103, 215, 215 | -0.035 (0.0386) | 0.197 (0.0267) | 0.237 (0.0267)
  FVC: Month 3, n=90, 197, 208 | -0.044 (0.0442) | 0.189 (0.0301) | 0.244 (0.0295)
  FVC: Month 6, n=79, 163, 178 | -0.002 (0.0478) | 0.206 (0.0330) | 0.237 (0.0320)
  FVC: Month 9, n=71, 142, 153 | -0.076 (0.0510) | 0.088 (0.0356) | 0.200 (0.0345)
  FVC: Month 12, n=66, 132, 143 | -0.039 (0.0491) | 0.155 (0.0343) | 0.213 (0.0333)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs were collected from on or after the date of the first dose of study drug to up to 1 day after the date of the last recorded dose of study drug (up to Study Week 52).
Description: On-treatment AEs and SAEs were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of randomized study drug.
Groups:
- Placebo: Participants received matching placebo once daily (QD) in the morning via a dry powder inhaler (DPI) for 52 weeks.ve
Arm/Group | Placebo | UMEC 125 µg | UMEC/VI 125/25 µg
Serious Adverse Events (participants affected / at risk) | 7/109 | 17/227 | 14/226
Other Adverse Events (participants affected / at risk) | 34/109 | 78/227 | 65/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=109) | UMEC 125 µg (N=227) | UMEC/VI 125/25 µg (N=226)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1
Myocardial fibrosis (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Rhythm idioventricular (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Clostridium test positive (Investigations) | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Skin graft (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=109) | UMEC 125 µg (N=227) | UMEC/VI 125/25 µg (N=226)
Nasopharyngitis (Infections and infestations) | 5 | 20 | 11
Sinusitis (Infections and infestations) | 3 | 6 | 8
Influenza (Infections and infestations) | 5 | 5 | 6
Upper respiratory tract infection (Infections and infestations) | 3 | 8 | 2
Headache (Nervous system disorders) | 9 | 25 | 20
Ventricular extrasystoles (Cardiac disorders) | 5 | 11 | 11
Extrasystoles (Cardiac disorders) | 4 | 10 | 10
Ventricular tachycardia (Cardiac disorders) | 4 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 9 | 10
Hypertension (Vascular disorders) | 5 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.